CLINICAL TRIAL: NCT06490042
Title: Children's Attitude Towards Helmet Use in Traffic.
Acronym: ChildHELMED
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Antoinette V. J. Rozeboom, Principal Investigator, Erasmus Medical Center
Other Study IDs: 12187
Record Dates: First submitted 2024-06-15; First posted 2024-07-08 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Helmets; Children; Behavior And Behavior Mechanism
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: The study group consists of children between 6 and 18 years presenting at the ED of the Erasmus Medical Centre (Erasmus MC) in Rotterdam after a bicycle accident between January 2017 and June 2024.
  Interventions: Behavioral: Questionnaire
- control group: The control group consists of children between 6 and 18 years in primary and secondary schools without a presentation at a ED after a bicycle accident in the past.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — A questionnaire about helmet use and attitude towards helmet use.

SUMMARY:
SUMMARY

Rationale:

Literature shows that helmet use is essential in the prevention of severe head injuries among children involved in bicycle accidents. However, helmet use in children remains low. Therefore, it is relevant to investigate the reason why helmet use among children is still low. In addition, it is unclear whether experiencing a serious bicycle accident influences helmet use and attitude towards helmet use among children.

Objectives:

Primary objective:

The aim of this study is to investigate the number of children using a bicycle helmet after visiting the emergency department (ED) following a bicycle accident compared to children who have not.

Secondary objective:

The secondary objective is to investigate children's attitude towards helmet use after visiting the ED following a bicycle accident compared to children who have not.

Other objectives:

To investigate the association between period of time after visiting the ED and attitude towards helmet use.

To investigate the association between type of injuries and attitude towards helmet use.

Study design: case control study

Study population:

The study group consists of children between 6 and 18 years presenting at the ED of the Erasmus Medical Centre (Erasmus MC) in Rotterdam after a bicycle accident between January 2017 and June 2024.

The control group consists of children between 6 and 18 years in primary and secondary schools without a presentation at a ED after a bicycle accident in the past.

Intervention:

A questionnaire about helmet use and attitude towards helmet use.

Main study parameters/endpoints:

The main study parameter is helmet use.

Secondary study parameters/endpoints:

The secondary parameter is attitude towards helmet use.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness:

A short, questionnaire will be administered. It takes around 10 minutes. There are no invasive interventions and thereby the risk and burden associated with participation in this study is considered low.

DETAILED DESCRIPTION:
This will be a case-control study consisting of two groups.

Hospital procedure Pediatric patients between 6 and 18 years old with a presentation at the ED of the Erasmus MC in Rotterdam after a bicycle accident between January 2017 and June 2024 will be registered into a database.

The researchers will contact these patients and ask them whether they're interested to participate in this study. The period of time between their accident and participation into the study must be at least 3 months.Patients that are interested will receive a letter at home containing detailed information about the study and a consent form. These patients have 4 weeks to carefully read everything and return the completed consent form by post. After this, a short, non-invasive questionnaire about helmet use and attitude towards helmet use will be administered.

Children aged 6 to 12 years will be be interviewed through a video call. In accordance with their parents/caregivers/representatives, an appointment will be scheduled to do this.Children aged 12 years and older will be asked to fill out an online questionnaire in their free time. They will receive it by email and so they can fill it out via their mobile phone, computer, tablet, etc. It takes around 10 minutes to fill out the questionnaire.

Information regarding the period of time between the visit to the ED and participation in the study; and injuries caused by the accident, as mentioned in other study parameter (8.1.3), will be collected from the electronic patient records (HIX).

School procedure To create a representative control group, potential participants are being selected based on the age and place of residence of the paediatric patients.

Therefore the researchers will contact primary and secondary schools and ask them whether they're interested to participate in this study. Schools that are interested will receive letters that the teachers can hand out to their students. These letters contain detailed information about the study and a consent form. These letters can only be given to students older than 6 years and younger than 18 years. Students have 4 weeks to carefully read everything an return a completed consent form to their teachers if they want to participate. After these weeks the researchers will visit the schools to collect the consent forms. After this, a short, non-invasive questionnaire about helmet use and attitude towards helmet use will be administered.

In case of primary school, children will be interviewed by the researchers. In accordance with the school and their teachers, an appointment will be scheduled to do this. In case of secondary schools, children will be asked to fill out an online questionnaire in their free time. They will receive it by email and so they can fill it out via their mobile phone, computer, tablet, etc. It takes around 10 minutes to fill out the questionnaire.

Reminder All participants who are asked to fill out an online questionnaire in their free time will receive an online reminder via email, in case they did not fill out their questionnaire after one month.

Informed consent procedures For children aged 6-12 years, informed consent must be obtained from their parents /caregivers/representatives. For children aged 12-16 years, informed consent must be obtained from both the parents/caregivers/representatives and the participants themselves. Children older than 16 can provide consent on their own. When informed consent is obtained, all participant will receive a copy at home.

Questionnaire To investigate attitude towards helmet use, a questionnaire is created based on the Health Belief Model (HBM). This model is widely used in research to investigate participant's behavior (35,36). This model defines the key factors that influence health behaviors as an individual's perceived threat to sickness or disease (perceived susceptibility), belief of consequences (perceived severity), potential positive benefits of action (perceived benefits), perceived barriers to action, exposure to factors that prompt action (cues to action) (37).

Perceived Susceptibility consists of 2 subscales. The first subscale is named Perceived Exemption from Harm and consists of 9 statements. Higher scores on these statements indicate more agreement with reasons for not needing a bicycle helmet in traffic. The second subscale is named Perceived Danger of Cycling and consists of 6 statements. Higher scores on these statements indicate more agreement with the perception that cycling can be dangerous.

Perceived Severity of Harm consists of 6 statements. Increased scores indicate a greater understanding of the potential severity of consequences associated with bicycling injury.

Perceived Benefits consists of 2 subscales. Emotional Benefits is the first one and consists of 5 statements. Higher scores reflect more agreement regarding the positive impact of helmet use on one's emotional status. Safety Benefits is the second subscale and consists of 4 statements. Higher scores suggest a stronger agreement that helmets can protect people against harm in a bicycle accident.

Perceived Barriers consist of 2 subscales. The first one is named Personal Vanity and Discomfort Barriers and consists of 10 statements. Higher scores indicate agreement with the idea that helmets are unattractive and uncomfortable. The second subscale is named Cost Barriers. Higher scores on these 5 statements indicate economic factors contributing to the decision to not wear a helmet.

Cues To Action consists of 5 subscales. The first one is named social circle. Higher scores on these 4 statements reflect a stronger agreement that participants receive support from friends and family to wear a helmet. The second subscale is Past Events. Higher scores on these 3 statements indicate that past bicycle accident related events influence helmet use. The third one is named Accessibility. Higher scores on these 3 statements suggest that a helmet is easily accessible. The fourth subscale is named Rules at Home and consists of 2 statements. Higher scores reflect agreement that parents/caregivers/representatives have or had rules about helmet use. The fifth subscale is named Rules at School and consists of 3 statements. Higher scores reflect agreement that their school focuses on traffic safety and helmet use.The last one is named Media. Higher scores on these 5 statements suggest that people receive information on bicycle helmets from various media sources.

Within the context of helmet use among cyclists, these elements may explain why some children choose to use a bicycle helmet while others do not.

ELIGIBILITY:
Inclusion criteria:

To be eligible for participation in this study, a patient must meet all of the following criteria:

* Presentation at the ED of the Erasmus MC in Rotterdam between January 2017 and June 2024 after a bicycle accident.
* Informed consent is obtained
* Aged between 6 and 18 years at moment of inclusion
* A maximum score on the Glasgow Coma Scale at the time the questionnaire is administered.
* Time between accident and questionnaire is at least 3 months

Inclusion criteria for the control group:

* Informed consent is obtained
* Using a bicycle
* Aged between 6 and 18 years at moment of inclusion

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation in this study:

* A non-bicycle accident (e.g. pedestrian, scooter, car)
* Being a bicycle passenger
* Linguistic barrier (unable to answer questions in Dutch or English)

Exclusion criteria for the control group:

* Presentation to any emergency department after a bicycle accident in the past.
* Being a bicycle passenger
* Linguistic barrier (unable to answer questions in Dutch or English)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — participants will be asked what their biological gender is.
Study Population: The study group consists of children between 6 and 18 years presenting at the ED of the Erasmus Medical Centre (Erasmus MC) in Rotterdam after a bicycle accident between January 2017 and June 2024.
  The control group consists of children between 6 and 18 years in primary and secondary schools without a presentation at a ED after a bicycle accident in the past.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Helmet use prevalence using a questionnaire | 6 months
  The number of children using a bicycle helmet after visiting the emergency department (ED) following a bicycle accident compared to children who have not.

SECONDARY OUTCOMES:
Helmet use attitude using a questionnaire | 6 months
  Children's attitude towards helmet use after visiting the ED following a bicycle accident compared to children who have not.

OTHER OUTCOMES:
Association between period of time post accident and attitude using a questionnaire and electronic patient files (EPF) | 6 months
  The association between period of time after visiting the ED and attitude towards helmet use.
Association between type of injury and attitude using a questionnaire and EPF | 6 months
  The association between type of injuries and attitude towards helmet use.

IPD SHARING:
Plan to Share IPD: No